CLINICAL TRIAL: NCT03309761
Title: Description of an Immune Activation Profile Linked to Insulin Resistance in Subjects Aged 55-69
Acronym: METACTIV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2016-02/PC-01; 2017-A01504-49 (Other: ANSM)
Record Dates: First submitted 2017-10-05; First posted 2017-10-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2019-09

CONDITIONS: Insulin Resistance; Metabolic Syndrome X
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 55-60
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — 6ml blood sample taken

SUMMARY:
The aim of the study is to describe an immune activation profile of people at risk of insulin resistance based on a wide range of markers which will allow easy identification of patients at risk.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been informed of the study, its objectives, constraints and the patient rights
* The patient must have given their free and informed consent and signed the consent form
* The patient is aged 55-69

Exclusion Criteria:

* The subject is participating in an interventional category 1 study
* The patient has participated in another category 1 interventional study in the last 3 months
* The patient is in a period of exclusion determined by a previous study
* The patient is under safeguard of justice or state guardianship
* The subject refuses to sign the consent
* The subject does not understand the information

Ages: 55 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers aged between 55-69
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Cluster of Differentiation 4 (CD4+) T cell subpopulations | Day 0
  immunosenescence; number/mm3
Cluster of Differentiation 8 (CD8+) T cell subpopulations | Day 0
  immunosenescence; number/mm3
B cell subpopulations | Day 0
  flow cytometry
Natural killer (NK) cell subpopulations | Day 0
  immunosenescence; number/mm3
sCD14 level | Day 0
  ng/ml, enzyme-linked immunosorbent assays (ELISA)
16 ribosomal ribonucleic acid (rRNA) levels | Day 0
  polymerase chain reaction (PCR); copies/µl
lipopolysaccharide (LPS)-binding protein level | Day 0
  ELISA; µg/mL
Intestinal Fatty Acid Binding Protein level | Day 0
  ELISA; pg/mL
Total cholesterol | Day 0
  mM/L
High Density Lipoprotein | Day 0
  mM/L
Low Density Lipoprotein | Day 0
  mM/L
fasting glycemia | Day 0
fasting insulinemia | Day 0
  mIU/L
γ-glutamyl transpeptidase level | Day 0
glutamic pyruvic transaminase | Day 0
hip circumference | Day 0
  cm
waist circumference | Day 0
  cm
minimal arterial tension | Day 0
  mmHg
maximal arterial tension | Day 0
  mmHg
Cluster of Differentiation 163 (CD163) level | Day 0
  ng/ml, enzyme-linked immunosorbent assays (ELISA)
soluble tumor necrosis factor-alpha receptor I (sTNFRI) level | Day 0
  ng/ml, enzyme-linked immunosorbent assays (ELISA)
soluble endothelial protein C Receptro (sEPCR) level | Day 0
  ng/ml, enzyme-linked immunosorbent assays (ELISA)
tissue plasminogen activator (tPa) level | Day 0
  ng/ml, enzyme-linked immunosorbent assays (ELISA)

SECONDARY OUTCOMES:
Prevalence of insulin and metabolic syndrome | Day 0
  % subjects
Link between immune activation profile and other features of metabolic syndrome | Day 0
  logistic regression of individual markers
Immune activation linked to the profile | Day 0
  logistic regression

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Nimes, Nîmes
  - Centre d'examen de santé de la Sécurité Sociale de Nîmes, Nîmes

REFERENCES:
- [Result] Cezar R, Winter A, Desigaud D, Pastore M, Kundura L, Dupuy AM, Cognot C, Vincent T, Reynes C, Dunyach-Remy C, Lavigne JP, Sabatier R, Le Merre P, Maggia E, Corbeau P. Identification of distinct immune activation profiles in adult humans. Sci Rep. 2020 Nov 30;10(1):20824. doi: 10.1038/s41598-020-77707-6. PMID 33257766